CLINICAL TRIAL: NCT00992355
Title: Tobramycin 0.3% - Dexamethasone 0.1% Versus Tobramycin 0.3% - Dexamethasone 0.1% Plus Ketorolac Tromethamine 0.5% After Phacoemulsification Surgery. A Randomized Trial
Brief Title: Tobramycin-Dexamethasone Versus Tobramycin-Dexamethasone Plus Ketorolac After Phacoemulsification Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veroia General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGH-EYE01
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Cataract
Keywords: Cataract; Phacoemulsification; Treatment duration
MeSH Terms: conditions — Cataract | interventions — Tobramycin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobramycin 0.3% - Dexamethasone 0.1% (Active Comparator)
  Interventions: Drug: Tobramycin 0.3% - Dexamethasone 0.1%
- Tobramycin-Dexamethasone plus Ketorolac tromethamine (Active Comparator)
  Interventions: Drug: Tobramycin 0.3% - Dexamethasone 0.1% plus Ketorolac tromethamine 0.5%

INTERVENTIONS:
Drug: Tobramycin 0.3% - Dexamethasone 0.1%
  Arms: Tobramycin 0.3% - Dexamethasone 0.1%
Drug: Tobramycin 0.3% - Dexamethasone 0.1% plus Ketorolac tromethamine 0.5%
  Arms: Tobramycin-Dexamethasone plus Ketorolac tromethamine

SUMMARY:
This randomized controlled trial compares two regimens of topical therapy:

* tobramycin 0.3% - dexamethasone 0.1% (TobraDex®, Alcon), one drop four times/day
* combination of tobramycin 0.3% - dexamethasone 0.1% (TobraDex®, Alcon), one drop four times/day, plus Ketorolac tromethamine 0.5% (Acular®, Allergan), one drop three times/day. The topical treatment is administered for 28 days after phacoemulsification.

Patients are independently assessed by two ophthalmologists. On day 28, patients are evaluated for

* corneal edema
* conjunctival redness
* anterior chamber reaction. Moreover, the cases necessitating continuation of treatment are compared in the two groups on day 28 and 42.

ELIGIBILITY:
Inclusion Criteria:

* Phacoemulsification (due to cataract)
* Uneventful phacoemulsification surgery

Exclusion Criteria:

* Disruption of the anterior lens capsule
* Age-related macular degeneration
* Proliferative diabetic retinopathy
* Glaucoma

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Veroia General Hospital, Véroia, Greece